CLINICAL TRIAL: NCT05395221
Title: Making Resident Well-Being a (Virtual) Reality
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-01719
Record Dates: First submitted 2022-05-11; First posted 2022-05-27 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Assisted Meditation+ no intervention Group (Experimental): The first cohort will undergo weekly virtual reality guided meditations across a three-month rotation using the Guided Mediation Virtual Reality App available on the Oculus Quest 2 Virtual Reality system (Oculus, Menlo Park, CA). After completion of the three-month time span, residents will receive no intervention during the second three-month study period. . A post-study survey will be completed to assess for various parameters including residents desire for continuation of virtual reality guided meditation following completion of the survey, subjective value of virtual reality as a tool for burnout, and likeliness to recommend virtual reality guided meditation to a colleague.
  Interventions: Other: Guided Mediation Virtual Reality App
- No intervention + Virtual Reality Assisted Meditation group (Experimental): The second cohort will receive no intervention during the three-month block. After completion of the three-month time span, residents will take a follow-up MBI and then will cross over to the opposite group. After completion of the second three-month study period, an additional MBI will be completed by the residents.. A post-study survey will be completed to assess for various parameters including residents desire for continuation of virtual reality guided meditation following completion of the survey, subjective value of virtual reality as a tool for burnout, and likeliness to recommend virtual reality guided meditation to a colleague.
  Interventions: Other: Guided Mediation Virtual Reality App

INTERVENTIONS:
Other: Guided Mediation Virtual Reality App — Guided Meditation Virtual Reality App uses over 40 lush environments with 30 hours of guided meditations on Anxiety, Depression, Maternity, Resilience, Sleep, or Zen and 200 relaxing audio tracks using Virtual reality.

SUMMARY:
This study is a prospective cross-over trial examining the effect of virtual reality assisted meditation on resident reported well-being using validated scoring systems. The primary objective of this study is to evaluate the effectiveness of virtual reality guided meditation as a mechanism to improve plastic surgery resident well-being. The secondary objective is to assess resident likeliness to continue mindful meditation following completion of the study.

DETAILED DESCRIPTION:
All plastic surgery residents participating will spend three months with access to virtual reality assisted meditation and three months without access to this technology. Assessment scores will be taken before and after the first three month period, and then again following the second three month period.

ELIGIBILITY:
Inclusion Criteria:

* Current resident of NYU Langone Plastic Surgery (Academic Year 2022-2023)
* Consent to participation in the study

Exclusion Criteria:

* Any plastic surgery resident involved in conducting the study
* Any non-plastic surgery resident during the academic year 2022-2023
* Any plastic surgery resident choosing not to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Exhaustion as measured by Maslach Burnout Inventory (MBI) | Baseline, 3 month visit, 6 month visit
  Emotional exhaustion as measured by Maslach Burnout Inventory (MBI) before and after virtual reality guided meditations. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout.
  Higher scores in emotional exhaustion contribute to higher levels of burnout.
Change in Depersonalization as measured by Maslach Burnout Inventory (MBI) | Baseline, 3 month visit, 6 month visit
  Depersonalization as measured by Maslach Burnout Inventory (MBI) before and after virtual reality guided meditations. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Higher scores in depersonalization contribute to higher levels of burnout.
Change in personal accomplishment as measured by Maslach Burnout Inventory (MBI) | Baseline, 3 month visit, 6 month visit
  Personal accomplishment as measured by Maslach Burnout Inventory (MBI) before and after virtual reality guided meditations. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Lower scores in personal accomplishment are suggestive of a more severe degree of burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Thanik, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.